CLINICAL TRIAL: NCT06816290
Title: Being a Nursing Student in a Foreign Country: a Photovoice Study
Brief Title: Being a Nursing Student in a Foreign Country
Acronym: NURS-PHOTO
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Nursemin ÜNAL, Associate Prof., Ankara University
Other Study IDs: 2025/3
Record Dates: First submitted 2025-02-03; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Nursing Education; Cultural Adaptation; Education
Keywords: nursing students; photovoice; Cultural Adaptation; international education

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Photovoice: Photovoice is a participant-centered research method that allows participants to convey their experiences through visual data. This method is particularly used to understand social issues and the challenges individuals face. Participants take photos that they find meaningful related to the research topic and express their feelings, thoughts, and experiences through these images.
  In this study, the Photovoice method is used to visualize the experiences of being a nursing student in a foreign country. Participants share their cultural adaptation, educational processes, personal challenges, and overall life experiences through photos taken with their smartphones. The photos are then analyzed in-depth during face-to-face interviews with the participants, where they discuss the meaning of the photo, the reason for choosing it, and their personal experiences.
  Interventions: Other: This research uses a qualitative method called photovoice. Participants express their "experience of being a nursing student in a foreign country" through visuals and share their feelings and

INTERVENTIONS:
Other: This research uses a qualitative method called photovoice. Participants express their "experience of being a nursing student in a foreign country" through visuals and share their feelings and — Photovoice is a participant-centered research method that allows participants to convey their experiences through visual data. This method is particularly used to understand social issues and the challenges individuals face. Participants take photos that they find meaningful related to the research topic and express their feelings, thoughts, and experiences through these images.
  In this study, the Photovoice method is used to visualize the experiences of being a nursing student in a foreign country. Participants share their cultural adaptation, educational processes, personal challenges, and overall life experiences through photos taken with their smartphones. The photos are then analyzed in-depth during face-to-face interviews with the participants, where they discuss the meaning of the photo, the reason for choosing it, and their personal experiences.

SUMMARY:
Understanding the experiences and specific learning needs of international nursing students is crucial for the success of nursing education programs. Providing necessary support and adjustments to facilitate their adaptation process is essential. This study employs the Photovoice method, a qualitative research approach, allowing students to express their educational journey from their own perspectives. Through visual representation, they can communicate their experiences more effectively.

DETAILED DESCRIPTION:
In addition to the advantages of being a nursing student in a foreign country, students may face many challenges that affect both their personal and academic lives. The lack of social networks and support systems, combined with the stress of the educational process, can negatively impact academic success. Studying in a foreign language can be particularly challenging, especially in the early stages. Language barriers can cause difficulties in understanding both theoretical and practical aspects of nursing education, hindering interaction with peers, faculty, and health teams in clinical settings. This can slow down the learning process and lead to communication breakdowns. Adapting to a new culture can also be challenging for some students, leading to anxiety, loneliness, or depression. Additionally, studying abroad brings extra costs such as tuition fees, accommodation, transportation, and health insurance.

This research will use a qualitative research method called the photovoice technique. Students meeting the inclusion criteria will be informed about the study's purpose and method, and invited to participate. Students who agree to participate will first complete an Introductory Information Form. They will then be asked to submit three photos, taken with their smartphones, that they feel reflect their experiences of "living in a foreign country and being a nursing student" within a week. Before photo submission, participants will be provided with the photo-taking procedure and will be required to send their photos along with date and time information and brief descriptions. These photos will be stored by the responsible researcher with a code number on a personal computer, along with transcripts.

The second phase of data collection will involve scheduling interviews in a quiet and secure environment. During face-to-face interviews, open-ended questions from the Structured Individual Interview Form will be asked, and participants will be encouraged to express their feelings and thoughts about the photos they have taken. They will also be asked to choose one photo that best represents their experience of "living in a foreign country and being a nursing student," and explain why they chose it. The two assistant researchers will transcribe the participant's explanations directly during the interview for content analysis.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled in the English program of the Nursing Department at a university during the 2024-2025 academic year.
* Being registered in the nursing department with the international student quota.
* Having completed at least one semester of nursing education.
* Owning a smartphone capable of taking photos.
* Volunteering to participate in the study

Exclusion Criteria:

* Students who wish to withdraw from the study at any stage will not be included in the research.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population consists of foreign students enrolled in the English program of the Nursing Department at a private university.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2025-02-17 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Semi-structured Questions | Within 1 week after participating in the study and submitting the photos to the researcher
  The interview is supported by four semi-structured questions that encourage international students to express their experiences:
  What is it like to be a student at this school? What factors help you in your studies here? As an international student, what challenges do you face? Can you describe your experiences as a nursing student in a foreign country?

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Acavut, Assist. Prof., Study Chair — Ankara Medipol University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Merry L, Vissandjee B, Verville-Provencher K. Challenges, coping responses and supportive interventions for international and migrant students in academic nursing programs in major host countries: a scoping review with a gender lens. BMC Nurs. 2021 Sep 18;20(1):174. doi: 10.1186/s12912-021-00678-0. PMID 34537039
- [Background] Tanrıkulu, F., Öner, Ö., Gürcay, B., & Akgül, E. (2024). A Qualitative Study of Foreign Nursing Students' Experiences of Educational Process. Journal of Qualitative Research in Education, (39), 1-18. https://doi.org/10.14689/enad.39.1732
- [Background] Kol E, Arikan F, Arikan C, Yabarow F, Gunbayi I. Being an international nursing student in Turkey: A qualitative study. Perspect Psychiatr Care. 2021 Jan;57(1):66-72. doi: 10.1111/ppc.12525. Epub 2020 May 8. PMID 32383270